CLINICAL TRIAL: NCT03468478
Title: Comparison of the Efficacy and Safety of Sirolimus, Everolimus or Mycophenolate in Renal Transplant Recipients Receiving Induction With Anti-thymocyte Globulin, Tacrolimus and Prednisone
Brief Title: Comparison of the Efficacy and Safety of Sirolimus Versus Everolimus Versus Mycophenolate in Kidney Transplantation
Acronym: SEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, Principal Investigator, Hospital do Rim e Hipertensão
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRHipertensao
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Kidney Transplant Infection
MeSH Terms: interventions — Sirolimus; Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- sirolimus +tacrolimus (Experimental): Patients will receive initial dose of 0,05 mg/kg BID oftacrolimus to reach blood trough concentration between 3-5 ng/mL. Initial dose of sirolimus of 3mg once a day to reach blood trough concentration between 4-8 ng/mL.
  Interventions: Drug: Sirolimus
- everolimus +tacrolimus (Experimental): Patients will receive initial dose of 0,05 mg/kg BID de tacrolimus to reach blood trough concentration between 3-5 ng/mL. Initial dose of 1.5 mg BID of everolimus to reach blood trough concentration between 4-8 ng/mL.
  Interventions: Drug: Everolimus
- mycophenolate +tacrolimus (Active Comparator): Patients will receive initial dose of 0,1 mg/kg BID de tacrolimusto reach blood trough concentration between Fixed dose of mycophenolate (mycophenolate mofetil, 1 g BID or sodium mycophenolate, 720 mg BID).
  Interventions: Drug: Mycophenolic acid

INTERVENTIONS:
Drug: Sirolimus — sirolimus combined to reduced dose of tacrolimus
  Other Names: Rapamune
  Arms: sirolimus +tacrolimus
Drug: Everolimus — everolimus combined to reduced dose of tacrolimus
  Other Names: Certican
  Arms: everolimus +tacrolimus
Drug: Mycophenolic acid — Control arm: mycophenolate combined to regular tacrolimus
  Other Names: mycophenolate sodium
  Arms: mycophenolate +tacrolimus

SUMMARY:
This study was designed to compare 3 immunosuppression regimens: sirolimus and tacrolimus versus everolimus and tacrolimus versus mycophenolate and tacrolimus.

The primary outcome is the incidence of cytomegalovirus infection / disease, a relevant medical need in the absence of pharmacological prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients, adults of the first living or deceased donor kidney transplant;
2. Patients who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

1. Receptors with a medical history of nephrotic syndrome or focal and segmental glomerulosclerosis confirmed as the etiology of end-stage renal disease;
2. Receptors with poor understanding about chronic kidney disease and its treatment alternatives;
3. Receptors with early history of non compliance to treatment with immunosuppressive drugs;
4. Retransplantation;
5. Multi-organ recipients;
6. Recipients with BMI> 30 kg / m2;
7. KDPI> 80%;
8. Cold ischemia time greater than 24 hours;
9. Receptors with a percentage of anti-HLA antibodies above 50%, either class I or Class II;
10. Women of childbearing potential who do not undertake contraceptive methods (condoms or oral contraceptives).
11. Patients receiving immunosuppressive therapy prior to transplantation, except low dose of prednisone;
12. Patients with severe uncontrolled dyslipidemia;
13. Patients who have a known contraindication for administration of any of the immunosuppressive drugs provided for in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1209 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Rim, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toniato de Rezende Freschi J, Cristelli MP, Viana LA, Ficher KN, Nakamura MR, Proenca H, Dreige YC, de Marco R, de Lima MG, Foresto RD, Aguiar WF, Medina-Pestana J, Tedesco-Silva H. A Head-to-head Comparison of De Novo Sirolimus or Everolimus Plus Reduced-dose Tacrolimus in Kidney Transplant Recipients: A Prospective and Randomized Trial. Transplantation. 2024 Jan 1;108(1):261-275. doi: 10.1097/TP.0000000000004749. Epub 2023 Aug 1. PMID 37525373

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus +Tacrolimus | Everolimus +Tacrolimus | Mycophenolate +Tacrolimus
Started | 403 | 403 | 403
Completed | 86 | 90 | 90
Not Completed | 317 | 313 | 313

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus +Tacrolimus | Everolimus +Tacrolimus | Mycophenolate +Tacrolimus | Total
Number analyzed (Participants) | 86 | 90 | 90 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.35 (12.4) | 44.5 (14.76) | 44.15 (12.32) | 44.01 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 23 | 74
  Male | 64 | 61 | 67 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 16 | 32
  White | 61 | 56 | 60 | 177
  More than one race | 17 | 25 | 13 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 86 | 90 | 90 | 266

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Cytomegalovirus Infection or Disease
Description: Incidence of CMV infection/disease in three study groups (SRL, EVR anda MPS).
Time Frame: 12 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus +Tacrolimus | Everolimus +Tacrolimus | Mycophenolate +Tacrolimus
Number analyzed (Participants) | 86 | 90 | 90
Participants | 9 | 7 | 39

ADVERSE EVENTS:
Time Frame: 12 months
Description: Number of episodes of serious adverse events in each study group.
Arm/Group | Sirolimus +Tacrolimus | Everolimus +Tacrolimus | Mycophenolate +Tacrolimus
All-Cause Mortality (participants affected / at risk) | 2/86 | 1/90 | 3/90
Serious Adverse Events (participants affected / at risk) | 43/86 | 47/90 | 71/90
Other Adverse Events (participants affected / at risk) | 0/86 | 0/90 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus +Tacrolimus (N=86) | Everolimus +Tacrolimus (N=90) | Mycophenolate +Tacrolimus (N=90)
CMV infection (Infections and infestations) | 5 (5) | 6 (6) | 24 (25)
Dehiscence of the aponeurosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Acute graft dysfunction (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Renal artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Acute gastroenterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pyelonephritis (Renal and urinary disorders) | 4 (4) | 6 (6) | 5 (7)
Acute graft rejection (Renal and urinary disorders) | 7 (8) | 6 (6) | 5 (5)
Sepsis of pulmonary focus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Infection of the operative wound (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Sars-Cov-2 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Other (General disorders) | 19 (19) | 19 (21) | 28 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03468478/Prot_SAP_000.pdf